CLINICAL TRIAL: NCT01449071
Title: A Phase1/2, Randomized, Parallel-group, Double-Blind, Placebo-Controlled, Multicenter Study of the Safety and Pharmacokinetics of One 12 Week Treatment Cycle of Epratuzumab in Japanese Systemic Lupus Erythematosus (SLE) Subjects With Moderate to Severe Disease
Brief Title: Study Evaluating the Pharmacokinetics and Safety of Epratuzumab in Japanese Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SL0026
Record Dates: First submitted 2011-10-03; First posted 2011-10-07 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; Monoclonal antibody; B-cell immunotherapy; Epratuzumab
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — epratuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo Group (Placebo Comparator)
  Interventions: Biological: Placebo
- Epratuzumab 600 mg Group (Experimental)
  Interventions: Biological: Epratuzumab 600 mg
- Epratuzumab 100 mg Group (Experimental)
  Interventions: Biological: Epratuzumab 100 mg
- Epratuzumab 400 mg Group (Experimental)
  Interventions: Biological: Epratuzumab 400 mg
- Epratuzumab 1200 mg Group (Experimental)
  Interventions: Biological: Epratuzumab 1200 mg

INTERVENTIONS:
Biological: Placebo — Placebo infusions at study weeks 0, 1, 2, and 3.
  Arms: Placebo Group
Biological: Epratuzumab 400 mg — Epratuzumab 400 mg infusions at study weeks 0, and 2, and placebo infusion at study weeks 1 and 3.
  Arms: Epratuzumab 400 mg Group
Biological: Epratuzumab 1200 mg — Epratuzumab 1200 mg infusions at study weeks 0, and 2, and placebo infusion at study weeks 1 and 3.
  Arms: Epratuzumab 1200 mg Group
Biological: Epratuzumab 100 mg — Epratuzumab 100 mg infusions at study weeks 0, and 2, and placebo infusion at study weeks 1 and 3.
  Arms: Epratuzumab 100 mg Group
Biological: Epratuzumab 600 mg — Epratuzumab 600 mg infusions at study weeks 0, 1, 2, and 3.
  Arms: Epratuzumab 600 mg Group

SUMMARY:
The primary objective of the study is to evaluate the safety, tolerability and Pharmacokinetics (PK) of Epratuzumab in Japanese subjects with moderate to severe general SLE as add on to standard of care treatment during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Positive Anti-nuclear Antibody (ANA) at Screening (Visit 1)
* Current clinical diagnosis of Systemic Lupus Erythematosus (SLE) by American College of Rheumatology (ACR) criteria
* Active moderate to severe SLE activity as demonstrated by British Isles Lupus Assessment Group Index (BILAG)
* Active moderate to severe SLE disease as demonstrated by Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) total score on stable SLE treatment

Exclusion Criteria:

* Subjects who are breastfeeding, pregnant, or plan to become pregnant
* Subjects with active, severe SLE disease activity which involves the renal system and active, severe, neuropsychiatric SLE, defined as any neuropsychiatric element scoring BILAG level A
* Serious infections

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Area under the concentration time curve (AUC) | From baseline to 12 weeks
  AUC is defined as the area under the plot of plasma concentration of Epratuzumab against time after administration per subject.
  All measurements taken in the study (at administration day [day 0, 7, 14, 21] and the next four days of each administration day and week-4, 6, 8, 10, 12) are used to calculate AUC
Half-life (t1/2) | From baseline to 12 weeks
  Half-life is defined as the time taken for plasma concentrations of Epratuzumab to decline by one half per subject.
  All measurements taken in the study (at administration day [day 0, 7, 14, 21] and the next four days of each administration day and week-4, 6, 8, 10, 12) are used to calculate Half-life.
Maximum plasma Concentration (Cmax) | From Baseline to 12 weeks
  Plasma concentration of Epratuzumab for each pharmacokinetics parameter is measured at administration day (day 0, 7, 14, 21) and the next four days of each administration day and week-4, 6, 8, 10, 12.

SECONDARY OUTCOMES:
Incidence of anti-epratuzumab in plasma during administration over 12 weeks | Day 0 (initial administration day) and week 12 (end of the evaluation period)
  Blood drawing for anti- epratuzumab is carried out at initial administration day (day 0) and end of the evaluation period (week 12).

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (7):
- Japan (7):
  - 09, Fukuoka
  - 10, Fukuoka
  - 11, Fukuoka
  - 03, Kitakyushu
  - 01, Tokyo
  - 08, Tokyo
  - 12, Urayasu

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- [Derived] Tsuru T, Tanaka Y, Kishimoto M, Saito K, Yoshizawa S, Takasaki Y, Miyamura T, Niiro H, Morimoto S, Yamamoto J, Lledo-Garcia R, Shao J, Tatematsu S, Togo O, Koike T. Safety, pharmacokinetics, and pharmacodynamics of epratuzumab in Japanese patients with moderate-to-severe systemic lupus erythematosus: Results from a phase 1/2 randomized study. Mod Rheumatol. 2016;26(1):87-93. doi: 10.3109/14397595.2015.1079292. Epub 2015 Oct 19. PMID 26382733